CLINICAL TRIAL: NCT02903680
Title: Randomised Controlled Trial of Intravenous Dexamethasone to Prevent Relapse in the Treatment of Migraine in a Pediatric Emergency Department
Brief Title: RCT of IV Dexamethasone to Prevent Relapse in the Treatment of Migraine in a Paediatric ED
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Geneviève Tourigny-Ruel, Paediatric Emergency Physician, St. Justine's Hospital
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: 3662
Record Dates: First submitted 2016-01-04; First posted 2016-09-16 (Estimated); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Migraine
Keywords: Relapse Prevention; Children
MeSH Terms: conditions — Migraine Disorders | interventions — dexamethasone acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexamethasone group (Active Comparator): Dexamethasone 0.6 mg/kg IV (max 15 mg) before departure from the ED.
  Interventions: Drug: Dexamethasone group
- Placebo group (Placebo Comparator): The control group received a similar looking placebo (NaCl 0,9% IV) with the same volume.
  Interventions: Drug: Placebo group

INTERVENTIONS:
Drug: Dexamethasone group — The intervention of interest was the administration of dexamethasone 0.6 mg/kg IV (max 15 mg) before departure from the ED. The control group received a similar looking placebo (NaCl 0,9% IV) with the same volume.
  Other Names: Dexamethasone Acetate
  Arms: Dexamethasone group
Drug: Placebo group — Normal Saline 0,9% same volume
  Other Names: Normal Saline 0,9%
  Arms: Placebo group

SUMMARY:
Background: Headaches is one of the most common complaints of children in the ED and the treatment of pediatric migraine is largely based on extrapolation data from adult studies, limited pediatric trials, clinical experience and expert consensus. Despite the fact that dexamethasone has already been proven effective to reduce recurrence and is currently used in treating adults with migraine, no studies have looked at its use in the treatment of childhood migraine where relapse rate of about 50% are described in the 48h following successful treatment in the ED.

Objective: To examine the effectiveness of parenteral dexamethasone at preventing migraine recurrence in children and to study the risk factors for migraine relapse after discharge from the ED.

Methods: This a randomised, double-blind, placebo-controlled clinical trial among all children 8 to 17 years of age with a presumptive diagnosis of acute migraine and treated with a standardized protocol in the ED of the CHU Ste-Justine, a tertiary care pediatric hospital. After the parenteral administration of prochlorperazine or metoclopramide and diphenhydramine, the patients were randomised to receive either dexamethasone or a placebo. They were excluded from the intervention if they had a known allergy or absolute contraindications to receiving parenteral corticosteroids, if they were already on a corticosteroid regimen or if they did not respond to the initial abortive migraine therapy. All included patients were discharged on a 48-hour course of naproxen and with a headache diary to fill out and return. The primary outcome was the incidence of relapse in the 24-48h following discharge from ED. The secondary outcomes evaluated were the mean level of pain, the use of rescue medication after ED discharge, the return rate to the ED or the visit to a health care professional within 7 days including hospitalisation. The associated symptoms, the adverse events after parenteral corticosteroids and the risk factors for migraine relapse were also evaluated. A telephone follow-up was made to ensure the headache diary was completed and returned.

DETAILED DESCRIPTION:
Study design This was a randomised, double-blind, placebo-controlled clinical trial among children with a presumptive diagnosis of acute migraine in the ED. The study was approved by the institutional IRB and written informed assent and consent were obtained by the patient and a parent respectively, prior to enrolment.

Study setting All patients were treated in the ED of the CHU Ste-Justine, a tertiary care pediatric hospital with approximately 70 000 visits annually. For over 10 years, the members of this ED have been using a standardized protocol for the treatment of migraine. (7) This protocol suggests the administration of prochlorperazine and diphenhydramine, to decrease the rate of akathisia, if the patient is 8 years of age or more and presents with severe migraine (unable to perform normal activities) or status migrainosus (migraine that last more than 72 hours) to be followed by a few day-course of naproxen. Unfortunately, there was a shortage of prochlorperazine at the moment of the study, so a decision was made to use metoclopramide instead, another dopamine (D2) receptor antagonist known to be effective in the treatment of migraine in adults. (15) To minimize the impact of this research on the clinical management of patients, it was decided that migraine would be treated according to the standardized local protocol depending on the availability or not of prochlorperazine. This means that the treating physician did use the prochlorperazine protocol when possible and metoclopramide if not. This was accounted for in the randomization to insure balance distribution between groups. While using dual intervention decreased the homogeneity of the participants, it improved drastically our external validity.

Participants Inclusion criteria Patients were eligible if they were between 8 and 17 years of age and if they were presenting a diagnosis of acute migraine requiring treatment with an intravenous rescue therapy (either metoclopramide or prochlorperazine) because of the severity of the migraine according to the treating physician. In a prior study, the same group of pediatric emergency physicians had their migraine diagnosis confirmed by a pediatric neurologist in 64 of 68 patients.(16) Exclusion criteria Patients were excluded if they had a known allergy to any study drugs or a component or absolute contraindication to receiving corticosteroids such as: active untreated infections, systemic fungal infections, cerebral malaria, respiratory tuberculosis, hypertension, heart failure, renal or hepatic impairment, GI diseases, myasthenia gravis, diabetes, cataracts, glaucoma, seizure disorder, thyroid dysfunction, and thromboembolic tendencies. Also, patients who were already on corticosteroids were not eligible. Finally, patients who were initially recruited but who did not respond to the abortive migraine therapy (no modification in the pain level) were not randomized to receive the intervention or placebo. Information about these patients was kept but it was not included in the primary analysis.

Intervention/procedure As mentioned, all participants received a standardized treatment consisting of metoclopramide (0.5 mg/kg IV, maximum 10 mg, q 1h prn, maximum of 3 doses) or prochlorperazine (0.15 mg/kg IV over 2-3 minutes, maximum 10 mg) and diphenhydramine (0.5 mg/kg IV, maximum 25 mg). The intervention of interest was the administration of dexamethasone 0.6 mg/kg IV (max 24 mg) before departure from the ED. The control group received a similar looking placebo (NaCl 0,9% IV) with the same volume. All patients received a perfusion of D5% NaCl 0.9% at basal requirements during their stay in the ED and were discharged on a 48-hour course of naproxen (Naprosyn® 5 mg/kg/dose BID, max 500 mg) provided by our pharmacy.

Primary Outcome The primary outcome was the incidence of relapse following discharge from the ED and up to 48 hours after metoclopramide or prochlorperazine initial administration. Relapse was defined as either occurrence of any headache pain, regardless of its severity, after a pain free status, or any increase in the pain intensity in participants who left the ED with residual pain.

Secondary outcome The secondary outcomes was the mean level of pain using the VAS at 24 and 48 hours following the initial administration of metoclopramide or prochlorperazine, the use of any rescue medication after ED discharge, the return rate to the ED, or the visit to a health care professional within 7 days including hospitalization. Also, the associated symptoms (i.e. nausea, vomiting, photophobia and sonophobia), the adverse events after parenteral corticosteroids (heartburns, constipation, personality changes such as irritability, and sleeping problem) and the following risk factors for migraine relapse were evaluated: headache duration, past history of headache, presence of familial history of migraine, age, sex, rescue medication at home prior to ED visit, prophylaxis at home prior to ED visit, past history of neurology consultation, past history of CT scan, maximal pain intensity, pain intensity on arrival to ED and at discharge, duration of sleep in ED, quality of sleep in ED, treatment in ED, treatment at discharge, compliance with medication after discharge, time to return to school, time to return to normal activities, number of hour of sleep after discharge of ED, and quality of sleep at home after ED discharge.

Study protocol All eligible children for whom the treating physician prescribed the migraine protocol in the study setting were invited to participate in the study before administration of the first medication (either metoclopramide or prochlorperazine). Baseline demographic data, vital signs, characteristics and duration of the headache were recorded on a standard data form. Patients were asked to complete a standardized questionnaire during the ED stay with the help of their parents if needed. At time 0, prior to any treatment, patients rated their headache severity on a 100 mm visual analogue scale (VAS), on a 0 to 10 verbal numeric scale (VNS) and on a 4-point verbal numeric scale (VNS) as 0=no headache, 1=mild headache, 2=moderate headache or 3=severe headache. The participants were also asked to rate their headache on a 4-point functional disability scale as 0=no disability (i.e. able to function normally); 1=mild disability (i.e. able to perform all activities of daily living but with some difficulty); 2= moderate disability (i.e. unable to perform certain activities of daily living); 3= severe disability (i.e. unable to perform most to all activities of daily living, or requiring bed rest). The participants then received the standard abortive migraine therapy previously detailed. Patients rated their headache severity on the three scales previously mentioned 2 hours after the abortive medication was given or as soon as they woke up (if they fell asleep) and they were asked to report any associated symptoms (i.e. nausea, vomiting, photophobia and sonophobia) and adverse effects (severity, seriousness, time of onset and resolution). The same assessment was repeated at discharge. Patients were discharged according to the clinical decision of the ED physician. In the uncommon situation where a participant was hospitalized because he did not respond adequately to the abortive intervention, this patient was excluded from the study and was not offered the intervention. The rationale behind this procedure was that dexamethasone was given to decrease migraine recurrence but it could not be effective if the migraine did not regressed. Just before discharge and the removal of the intravenous access, the research nurse took the next available study package according to the status of the patient (absence or presence of residual pain at discharge and abortive medication used) and administered the intervention, either the study drug or the placebo. All patients were discharged on a 48-hour course of naproxen provided by our pharmacy to facilitate compliance at a dosage of 5 mg/kg twice a day for 48 hours. The participants were also given a headache diary to fill out and a stamped envelop with the standardized questionnaire used by the research assistant for follow up in case the phone interview would not happen. The participants were instructed to answer the questions of the diary once a day for the first 48 hours after discharge and then on day 4 and 7 and to then return the diary in the stamped envelop. To facilitate compliance with the headache diary, patients were contacted by telephone at 24-48 hours and one week later to remind them to complete and return the diary and they were also asked the same questions by the research assistant on the phone.

Randomization and blinding The hospital pharmacist created the randomization table using computer generated sequence using block randomization of variable sizes. Stratification was performed according to the absence or presence of pain at discharge and also depending on the abortive medication used (prochlorperazine or metochlopramide). The pharmacist coded the study medications in advance. Either dexamethasone (10 mg/mL) or normal saline (placebo) was placed into each respective syringe and labeled with a code number. Once consent for study enrolment was obtained, the next consecutive study package was used. Blinding was assured by dexamethasone and placebo having the same appearance and being administered in the same volume.

Compliance and quality control Because the intervention was limited to a single dose of intravenous medication, compliance was almost perfect. However, we did ensure that the dose was effectively given to the participants according to their charts. Several precautions were taken in order to minimize potential biases. A screening log was maintained to record the number of patients screened, excluded, missed, or not randomized for any other reason. The diagnosis and reason for exclusion (ineligible or refused patients) was recorded in order to help us in detecting any selection bias. We also implemented a number of study manoeuvres aimed at minimizing measurement biases, including (a) designation of a research pharmacist (not a team member) to prepare the medications according to the randomization list, and (b) documenting the use of any major co-intervention, such as the use of other analgesia.

Statistical analysis All data were entered in an Excel database (Microsoft Inc., Richmond, WA) and analyzed with SPSS v17 software (SPSS Inc., Chicago, Illinois). To assess balance across arms, baseline demographic (i.e. gender, age) and clinical data of patients were compared between arms. In the very unlikely event that a substantial imbalance is found, additional analyses, in addition to the one proposed below, were carried out to assess the potential confounding effects of this imbalance. The primary analysis was performed among all study participants who received the study medication using an intention-to-treat principle. This was the comparison of the proportion of relapse in the 48 hours following intervention between the 2 groups using chi-square analysis. A secondary analysis compared relapse proportion at one week. Another secondary analysis used a student t-test to compare mean VAS for pain at 24 hours, 48 hours and 7 days following intervention. Finally, use of rescue medication, unplanned visit to a healthcare setting and side effects were compared using a chi-square statistics.

Sample size requirement A previous study done in a pediatric emergency department had reported that approximately 50% of children successfully treated for migraine in our study setting had a relapse in the following 48 hours.(7) Based on this, the minimal clinically significant difference was defined a-priori by our group of pediatric emergency physicians to be a decrease of that relapse rate to 25%. Assuming these numbers, a total of 58 patients were required in each group for a power of 0.80 with an alpha of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* presenting a diagnosis of acute migraine
* requiring treatment with an intravenous rescue therapy (either metoclopramide or prochlorperazine) because of the severity of the migraine according to the treating physician.

Exclusion Criteria:

* known allergy to any study drugs or a component
* absolute contraindication to receiving corticosteroids such as: active untreated infections, systemic fungal infections, cerebral malaria, respiratory tuberculosis, hypertension, heart failure, renal or hepatic impairment, GI diseases, myasthenia gravis, diabetes, cataracts, glaucoma, seizure disorder, thyroid dysfunction, and thromboembolic tendencies
* patients who were already on corticosteroids
* patients who were initially recruited but who did not respond to the abortive migraine therapy (no modification in the pain level) were not randomized to receive the intervention or placebo.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 116 (Estimated)
Dates: Start 2014-05 (Actual); Primary Completion 2025-03-03 (Actual); Study Completion 2025-03-03 (Actual)

PRIMARY OUTCOMES:
incidence of relapse following discharge from the ED | 7 days
  by questionnaire

SECONDARY OUTCOMES:
mean level of pain | at 24 and 48h post intervention
  using the visual analog scale (VAS)
associated symptoms (i.e. nausea, vomiting, photophobia and sonophobia), | 7 days
  by questionnaire
adverse events after parenteral corticosteroids | 7 days
  by questionnaire (heartburns, constipation, personality changes such as irritability, and sleeping problem ad 7 days
risk factors for migraine relapse | 7 days
  questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Benoit Bailey, MD, Principal Investigator — Ste-Justine's Hospital
Locations (1):
- CHU Sainte Justine, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No